CLINICAL TRIAL: NCT03577795
Title: A Prospective Cohort Study of Asthma and COPD Overlap in Japanese COPD Patients Using the Diagnostic Criteria of The Japanese Respiratory Society
Acronym: ACO-Registry
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Linical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00005
Record Dates: First submitted 2018-05-23; First posted 2018-07-05 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD, ACO, RWE
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicentered and non-interventional prospective cohort study. Study centers shall be the institutions where the examinations, adopted in the ACO diagnostic criteria9) from The Japanese Respiratory Society, are performed at least once a year as a part of their regular practice. Physicians participating in the study will consecutively register by means of central registration outpatients who have the characteristics of COPD in the ACO diagnostic criteria9) from The Japanese Respiratory Society, and who have been confirmed to satisfy the inclusion criteria whereas not violating the exclusion criteria.

DETAILED DESCRIPTION:
This study is a multicentered and non-interventional prospective cohort study. Study centers shall be the institutions where the examinations, adopted in the ACO diagnostic criteria9) from The Japanese Respiratory Society, are performed at least once a year as a part of their regular practice. Physicians participating in the study will consecutively register by means of central registration outpatients who have the characteristics of COPD in the ACO diagnostic criteria9) from The Japanese Respiratory Society, and who have been confirmed to satisfy the inclusion criteria whereas not violating the exclusion criteria. The physicians will collect data including the patients' results from medical examinations by using the ACO diagnostic criteria, at each time point (on the registration, after 1 year, and after 2 years). Electronic case report forms completed by participating physicians and questionnaires completed by patients will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from whom written consent to participate in this study has been obtained
2. Patients ≥40 years old
3. Patients with FEV1/FVC ratio <70% after bronchodilator inhalation within the past year or on the registrationa
4. Patients who satisfy any one of the following items:

1) Smoking history (≥10 pack-years) or comparable air pollution exposure on the registrationa 2) Presence of the low attenuation area on chest CT demonstrating emphysematous alteration within the past year or on the registration a,b, 3) Impaired pulmonary diffusing capacity (%DLCO <80% or %DLCO/VA <80%) within the past year or on the registrationa 4) Patients deemed capable of visiting their study center in Japan at least once a year on an outpatient basis

Exclusion Criteria:

1. Patients who participated in other interventional studies such as clinical trial within the last 8 weeks.
2. Patients who are unsuitable for their enrollment in this study, judged by the participating physician, because they cannot comply with the procedures, restrictions, and requirements of this study (e.g., patients with dementia).
3. Patients with exacerbationsa of COPD or asthma within the last 8 weeks. a COPD exacerbation: State of increased shortness of breathing, increased cough and sputum, and occurrence or exacerbation of chest discomfort that requires a change of treatment during the stable phase. However, exacerbation preceded by other disorders (e.g., heart failure, pneumothorax, pulmonary thromboembolism) is excluded.

   Asthma exacerbation: Occurrence of paroxysmal/variable cough/sputum/wheezing/dyspnea caused by various factors including respiratory infection.
4. Patients carrying following disorders that should be distinguished from COPD or asthma:

Diffuse panbronchiolitis, congenital sinobronchial syndrome, occlusive panbronchiolitis, bronchiectasis, pulmonary tuberculosis, pneumoconiosis, lymphangioleiomyomatosis, congestive heart failure, interstitial lung disease, lung cancer, laryngitis, epiglottitis, vocal cord dysfunction, intratracheal tumor, airway foreign substance, tracheomalacia, bronchial tuberculosis, pulmonary thromboembolism, cough induced by drug such as angiotensin-converting enzyme inhibitor, spontaneous pneumothorax, hyperventilation syndrome, psychogenic cough

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients should be 40 years old or older who satisfy the characteristics of COPD from The Japanese Respiratory Society's ACO diagnostic criteria within the past years or on the registration as well as who can regularly visit their study center in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Prevalance of ACO | 2 years
  1. Proportion of patients diagnosed with ACO at least once at the time of registration, 1 year later, and 2 years later among all registered patients
  2. The number and proportion of ACO patients and non-ACO patients at the time of registration among patients who have data required for the diagnosis of ACO at the time of registration

CONTACTS AND LOCATIONS:
Overall Officials: Masakazu Ichinose, Professor, Study Chair — Tohoku University School of Medicine
Locations (1):
- Tohoku University School of Medicine, Sendai, Miyagi, Japan

REFERENCES:
- [Derived] Hashimoto S, Sorimachi R, Makita N, Tashiro N, Sugaya S, Arita Y, Ichinose M. Real-World Status of Medical Care and Treatment of Chronic Obstructive Pulmonary Disease by Respiratory Specialists in Japan. Adv Ther. 2022 Oct;39(10):4509-4521. doi: 10.1007/s12325-022-02167-5. Epub 2022 Jun 29. PMID 35767123
- [Derived] Hashimoto S, Sorimachi R, Jinnai T, Ichinose M. Asthma and Chronic Obstructive Pulmonary Disease Overlap According to the Japanese Respiratory Society Diagnostic Criteria: The Prospective, Observational ACO Japan Cohort Study. Adv Ther. 2021 Feb;38(2):1168-1184. doi: 10.1007/s12325-020-01573-x. Epub 2020 Dec 23. PMID 33355907
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00005&attachmentIdentifier=69af77e1-081f-4a34-8021-f959319d7bb0&fileName=ASZ006_CSR_synopsis_ver.1.pdf&versionIdentifier=